CLINICAL TRIAL: NCT03866460
Title: Determination of Hearing Status in Children Receiving Intra-Arterial Carboplatin for Intraocular Retinoblastoma
Brief Title: Determining Whether Intra-Arterial Carboplatin Causes Hearing Loss in Children
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-529
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Intraocular Retinoblastoma; Hearing Loss
Keywords: Hearing Status; 18-529
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hearing evaluation DPOAE: Post IA hearing evaluation will be allowed up until 9 months after IA completion (or roughly one year from initiation of treatment). After completion of standard treatment for RB that included IA carboplatin.
  Interventions: Diagnostic Test: Distortion product otoacoustic emission measurement (DPOAE)

INTERVENTIONS:
Diagnostic Test: Distortion product otoacoustic emission measurement (DPOAE) — Hearing will be measured at baseline and 3-9 months after completion of treatment with IA carboplatin chemotherapy.

SUMMARY:
The purpose of this study is to find out how often hearing loss occurs in patients with retinoblastoma after receiving treatment with intra-arterial carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent indicating awareness of the investigational nature of the protocol.
* Children with RB aged 3 months and older who are scheduled to receive their first dose of IA carboplatin chemotherapy.

  * Retinoblastoma is rarely seen in children over 8 years old, however we will not include an upper age range so as not to exclude any possible participants

Exclusion Criteria:

* Children with known and documented preexisting hearing loss.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients will be identified from the retinoblastoma clinic when the treatment plan includes IA carboplatin chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Estimate the incidence of hearing loss | 1 year
  will be defined as a >10 db loss from baseline in any frequency, based on the lower threshold of the American Speech and Hearing Associations (ASHA) hearing change criteria. For children unable to cooperate for an audiogram, the DPOAE will be the primary measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elizabeth Davis, MSN, RN, AOCNS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm